CLINICAL TRIAL: NCT02566408
Title: Attitudes, Beliefs and Preferences of Older Breast Cancer Survivors Towards Physical Activity
Brief Title: Attitudes, Beliefs, and Preferences of Older Stage I-III Breast Cancer Survivors Towards Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE5115; NCI-2015-01052 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE 5115 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2015-09-29; First posted 2015-10-02 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Cancer Survivor; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (interview about KAPs towards PA) (Experimental): Participants undergo a 2-hour one-on-one interview and answer survey questions about their beliefs, attitudes, and preferences (KAPs) towards physical activity (PA). Ten topics will be used to explore older women's attitudes toward PA. Six topics will also be used to explore ethnic-specific and culture-specific contexts that surround older women's participation in PA.
  REFINEMENT OF THE PA INTERVENTION: Approximately 1-2 months after the conclusion of interviews, participants are invited to a joint session and presented with results of analyzed data. Participants are asked to review results and themes identified from interviews, and to concur whether conclusions capture their KAPs. Through this process a set of preferences that is agreed upon by all as most critical for enhancing PA participation, adherence, and retention will be identified.
  Interventions: Other: One-on-one interview; Other: Survey Questions

INTERVENTIONS:
Other: One-on-one interview — Undergo one-on-one interview about KAPs towards PA
Other: Survey Questions — Complete survey

SUMMARY:
This clinical trial studies the attitudes, beliefs, and preferences of older stage I-III breast cancer survivors towards physical activity. Studies have shown that older African-American and women of lower socioeconomic status are more likely than their Caucasian counterparts and women of higher socioeconomic status to have functional disability at the time of a new breast cancer diagnosis. Functional disability is the inability to independently complete activities of daily living and increases health care costs and deaths. The poor health status of older African-Americans with breast cancer has been suggested to diminish the long-term benefits from cancer treatment, resulting in older African-American women more likely to die from breast cancer compared to Caucasians. Questionnaires that measure the attitudes, beliefs, and preferences of older breast cancer survivors may lead to the development of an intervention that increases physical activity, improves functional and health status, and improves breast cancer treatment benefits translating to improved survival among older breast cancer survivors in general, and in particular among older African-American and lower socioeconomic status women with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess physical activity beliefs, attitudes and preferences (KAPs) of breast cancer (BCa) survivors to inform the development of a physical activity (PA) intervention that will foster initial enrollment and sustained participation, particularly for African American (AA) and socioeconomic status (SES)-disadvantaged BCa survivors.

OUTLINE:

INTERVIEWS AND GROUP DISCUSSION: Participants undergo a 2-hour one-on-one interview about their KAPs towards PA. Ten topics will be used to explore older women's attitudes toward PA: (a) terminology used to describe PA; (b) meaning of PA to older women; (c) usual PA during daily life; (d) perceived influences and benefits of PA on body and mind; (e) recent changes in PA and their influences on women's daily life; (f) facilitators and barriers to older women's participation in PA; (g) preferences for PA in general and specific types of PA; (h) age-related differences in attitudes toward PA; (i) ethnic differences in attitudes toward PA; (i) SES-related differences in attitudes toward PA; and (j) overall feeling about PA. Six topics will also be used to explore ethnic-specific and culture-specific contexts that surround older women's participation in PA: (a) older women's daily life schedules, and hardships and sufferings in daily lives; (b) culturally unique aspects of women's daily lives; (c) age-related difficulties and advantages in daily lives influencing older women's participation in PA; (d) ethnicity-related, cultural-related and SES-related difficulties and advantages in daily lives influencing women's participation in PA; (f) culturally available support for PA and women's preferences for support; and (g) older women's preferences for PA promotion programs.

REFINEMENT OF THE PA INTERVENTION: Approximately 1-2 months after the conclusion of interviews, participants are invited to a joint session and presented with results of analyzed data. Participants are asked to review results and themes identified from interviews, and to concur whether conclusions capture their KAPs. Through this process a set of preferences that is agreed upon by all as most critical for enhancing PA participation, adherence, and retention will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed breast cancer
* Stage I-III
* Patients who have completed treatment for breast cancer and are within two years of treatment completion (primary surgery, chemotherapy or radiation therapy), whichever was received last; hormonal therapy and targeted therapies in the adjuvant setting are allowed
* African-Americans and non-Hispanic Whites

Exclusion Criteria:

* Stage IV breast cancer
* Patients with end-stage disease, severe dementia and/or life expectancy of less than one year
* Inability to understand English
* Inability to provide informed consent

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-10-14 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2016-10-01 (Actual)

PRIMARY OUTCOMES:
Qualitative analysis of in-depth interviews to identify features which foster initial enrollment of African Americans and Socioeconomic Status disadvantaged breast cancer survivors in breast cancer studies | 6 months
  Features of the physical activity program that are important to the initial enrollment of older breast cancer survivors, particularly African American and Socioeconomic Status disadvantaged breast cancer survivors. These features will be analyzed using descriptive statistics. Examining the data by groups will further refine understanding of the emergent themes. Discussion of the findings and suggestions for interpretation will be used to guide subsequent analyses to more fully understand the themes and patterns among the themes.
Qualitative analysis of in-depth interviews to identify attitudes towards physical activity. | 6 months
  Identification of attitudes of survivors toward physical activity will be analyzed using descriptive statistics. Examining the data by groups will further refine understanding of the emergent themes. Discussion of the findings and suggestions for interpretation will be used to guide subsequent analyses to more fully understand the themes and patterns among the themes.
Qualitative analysis of in-depth interviews to identify attitudes towards the physical activity program. | 6 months
  Identification of attitudes of survivors toward the physical activity program will be analyzed using descriptive statistics. Examining the data by groups will further refine understanding of the emergent themes. Discussion of the findings and suggestions for interpretation will be used to guide subsequent analyses to more fully understand the themes and patterns among the themes.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Owusu, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States